CLINICAL TRIAL: NCT02991612
Title: Efficacy of Rafiximin in Patients With Cirrhotic Gastroesophageal Variceal Hemorrhage: A Single-center Pilot Study
Brief Title: Rifaximin in Patients With Gastroesophageal Variceal Bleeding
Acronym: RFXM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-CSY-RFXM
Record Dates: First submitted 2016-12-10; First posted 2016-12-13 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cirrhosis; Esophageal and Gastric Varices; Gastrointestinal Hemorrhage
MeSH Terms: conditions — Fibrosis; Esophageal and Gastric Varices; Gastrointestinal Hemorrhage | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rifaximin Treatment Group (Experimental): Rifaximin 400mg bid for 2 months,
  Interventions: Drug: Rifaximin
- Control Group (No Intervention): Receive routine endoscopic treatment without having rifaximin for 2 months

INTERVENTIONS:
Drug: Rifaximin — Patients receive Rifaximin 400mg bid for 2 months
  Other Names: XIFAXAN
  Arms: Rifaximin Treatment Group

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of Rifaximin in the treatment of cirrhotic gastroesophageal variceal bleeding.

DETAILED DESCRIPTION:
Gastroesophageal variceal bleeding is the most common and life-threatening condition in patients with portal hypertension, which are susceptibility to bacterial infection.

However, the prophylaxis use of antibiotics remained uncertain and lack of high level evidences.

ELIGIBILITY:
Inclusion Criteria:

* 18 y.o. ≤age≤75 y.o.;
* Cirrhotic gastroesophageal variceal bleeding underwent endoscopic treatment (include esophageal varices ligation, endoscopic injection sclerosis and gastric N- butyl-cyanoacrylate injection).

Exclusion Criteria:

* age <18 y.o. or age > 75 y.o.;
* Never had the variceal bleeding episode before;
* Do not have endoscopic treatment;
* Combined with other malignant tumors (not exclude patients with hepatocellular carcinoma who don't need treatment at the moment);
* Known infection after endoscopic treatment (Fever, microbial cultures positive, et al.)
* Massive ascites or combined with other high-risk factors that require prophylaxis use of antibiotics.
* Acute variceal bleeding within 5 days.
* Refuse to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of all clinical adverse events | 8 weeks
  The occurrence of rebleeding, ascites fluid infection, hepatorenal syndrome, hepatopulmonary syndrome, portal vein thrombosis, or death in 8 weeks

SECONDARY OUTCOMES:
Changes of portal vein thrombosis | 2 months
  complete or partial recanalization of thrombosis
Changes of intestinal flora | 2 months
  Metagenomics sequencing
The changes of serum level of cytokines | 8 weeks
  Cytokines including TNF-α, IL-1β, IL-2R, IL-6 and IL-10, etc

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao CHEN, M.D., Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Huang XQ, Ai YJ, Li F, Ye ST, Wang JH, Zhang R, Zhang W, Zhu YL, Chen SY. Impact of rifaximin on cirrhosis complications and gastric microbiota in patients with gastroesophageal variceal bleeding: A pilot randomized controlled trial. J Dig Dis. 2024 Aug;25(8):504-516. doi: 10.1111/1751-2980.13314. PMID 39443081
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180